CLINICAL TRIAL: NCT03091478
Title: Pembrolizumab in Patients With Leptomeningeal Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J16156; IRB00116423 (Other: JHM IRB)
Record Dates: First submitted 2017-01-03; First posted 2017-03-27 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Patients With Leptomeningeal Disease
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab 200 mg (Experimental): Pembrolizumab 200 mg every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg every 3 weeks
  Other Names: Keytruda

SUMMARY:
This is an open-label phase II study of pembrolizumab in patients with advanced solid tumors with leptomeningeal carcinomatosis (LMD). Approximately 18 subjects in this study will receive pembrolizumab at a dose of 200mg intravenously (IV) every 3 weeks (Q3W) for 4 doses.

DETAILED DESCRIPTION:
This is an open-label phase II study of pembrolizumab in patients with advanced solid tumors with leptomeningeal carcinomatosis (LMD). Patients may have received any number of prior therapies for their respective solid tumors, but must not have received prior anti-PD-1 therapy and developed progressive disease. Approximately 18 subjects in this study will receive pembrolizumab at a dose of 200mg intravenously (IV) every 3 weeks (Q3W) for 4 doses. In patients who derive clinical benefit from therapy, pembrolizumab may be continued until documented disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdrawal of consent, noncompliance with trial treatment or procedure requirements, or for administrative reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial.
2. 18 years of age on day of signing informed consent.
3. Histologically or cytologically confirmed solid tumor malignancy.
4. Cytologically confirmed LMD or radiologically detectable LMD defined as either/or:

   A measurable lesion on contrast-enhanced MRI of either the Brain or Total Spine greater than 3mm that has not been radiated within the last 3 months prior to commencement of study therapy.

   Positive cerebrospinal fluid (CSF) cytology
5. Patients may be newly diagnosed or have received any number of lines of prior anti cancer therapy. However, patients are required to have received available therapies for their primary disease, as deemed appropriate by the treating investigator.
6. Non escalating steroid requirement at the time of consent and study drug initiation for the treatment of central nervous system (CNS) symptoms.
7. Local radiation therapy (RT) is allowed as needed to manage symptoms appropriately, as long as there remains a measurable lesion in the CNS.
8. Whole brain RT may be used, without a pre-defined washout period, prior to commencement of study therapy if the lesion that has been radiated is not the sole measurable lesion, or the patient is eligible based on positive CSF cytology.
9. Patients may continue therapy with a targeted agent if CNS disease developed while receiving the agent, and for defined regimens that have been deemed safe when combined with anti PD 1 therapy.
10. Be willing to provide tissue from an archival tissue specimen in selected patients, where available.
11. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
12. Demonstrate adequate organ function as defined in Table 3, all screening labs should be performed within 10 days of treatment initiation.

    Table 3.
13. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Female subjects of childbearing potential (Section 4.8.2) must be willing to use an adequate method of contraception as outlined in Section 4.8.2 Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
15. Male subjects of childbearing potential (Section 4.8.2) must agree to use an adequate method of contraception as outlined in Section 4.8.2 Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks or 5 half lives of the first dose of treatment, whichever is shorter.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy other than pre specified allowed agents detailed in section 4.2.6, or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. All major surgery including prior surgery to the brain within 3 weeks of commencement of study therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Subjects with previously treated brain metastases may participate provided they are not using escalating steroids for brain metastases at the time of trial consent and study drug initiation, and there remains a measurable lesion in the CNS, as per section 4.2.6.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Prior disease progression on anti-PD-1 therapy
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (HCV) (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy.
20. Contraindication to MRI.
21. Patients with a condition related to their cancer or leptomeningeal disease requiring urgent intervention that has not been clinically managed or stabilized prior to the time of consent.
22. Brain metastases with risk of mass effect that would contraindicate lumbar puncture, as detailed in section 6.1.2.8.3.
23. Live vaccines within 30 days prior to the first dose of trial treatment. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarushka Naidoo, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Naidoo J, Schreck KC, Fu W, Hu C, Carvajal-Gonzalez A, Connolly RM, Santa-Maria CA, Lipson EJ, Holdhoff M, Forde PM, Douville C, Riemer J, Barnes A, Redmond KJ, Kleinberg L, Page B, Aygun N, Kinzler KW, Papadopoulos N, Bettegowda C, Venkatesan A, Brahmer JR, Grossman SA. Pembrolizumab for patients with leptomeningeal metastasis from solid tumors: efficacy, safety, and cerebrospinal fluid biomarkers. J Immunother Cancer. 2021 Aug;9(8):e002473. doi: 10.1136/jitc-2021-002473. PMID 34380662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Eligible patients who receive at least one dose of pembrolizumab.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 13
Participants
  Complete Response | 2
  Partial Response | 1
  Stable Disease | 2
  Progressive Disease | 8

2. Secondary Outcome: CNS Progression-free Survival in Patients With LMD From Solid Tumors Receiving Pembrolizumab
Description: To determine whether pembrolizumab administered in patients with Leptomeningeal disease (LMD) from solid tumors improves central nervous system (CNS) progression-free survival (PFS).
Time Frame: From the date of study entry until date of death from any cause, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 13
Months | 2.9 [1.3 to NA] — The upper bound of the confidence interval was not reached.

3. Secondary Outcome: Overall Survival in Patients With LMD From Solid Tumors Receiving Pembrolizumab
Description: To determine whether pembrolizumab administered in patients with LMD from solid tumors improves overall survival (OS).
Time Frame: From the date of study entry until date of death from any cause, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 13
Months | 4.9 [3.7 to NA] — The upper bound of the confidence interval was not reached.

ADVERSE EVENTS:
Time Frame: For the time period beginning at treatment allocation/registration through 90 days following cessation of treatment, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier.
Arm/Group | Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 9/13
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=13)
Nausea (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Weakness, Lower Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Thrombolic Event- PE (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=13)
Hypothyroidism (Endocrine disorders) | 1 (1)
Anisocoria (Eye disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (2)
Dry Eye (Eye disorders) | 1 (1)
Twitching Eyelid (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 5 (7)
Face Edema (General disorders) | 1 (1)
Edema Limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 6 (10)
Fever (General disorders) | 1 (1)
Infusion Related Reaction (General disorders) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2)
Creatinine Increased (Investigations) | 1 (1)
Weight Loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (7)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (16)
Precancerious Cells from Scalp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Cerebrospinal fuild leakage (Nervous system disorders) | 1 (1)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Concentration Impairment (Nervous system disorders) | 1 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysphagia (Nervous system disorders) | 1 (1)
Edema Cerebral (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (8)
Lethargy (Nervous system disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Delusions (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (4)
Minimal Redness at site of LP (General disorders) | 1 (1)
Left cheek lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (6)
Hypotension (Vascular disorders) | 1 (1)
Left supine craniotomy (Surgical and medical procedures) | 1 (1)
Confusion (Nervous system disorders) | 2 (3)
Dysarthria (Nervous system disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03091478/Prot_SAP_000.pdf